CLINICAL TRIAL: NCT00956566
Title: Randomized Parallel Group Comparison on the Influence of a Low Carbohydrate and a Low Fat Hypocaloric 6 Months Diet on Body Weight Reduction, Metabolic and Cardiovascular Variables in Obese Healthy Women and Men.
Brief Title: Comparison of Low Fat and Low Carbohydrate Diets With Respect to Weight Loss and Metabolic Effects
Acronym: B-SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jens Jordan, Prof. Dr. med., Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-SMART
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low fat hypocaloric diet (Active Comparator)
  Interventions: Behavioral: dietary intervention
- Low carbohydrate hypocaloric diet (Active Comparator)
  Interventions: Behavioral: dietary intervention

INTERVENTIONS:
Behavioral: dietary intervention — dietary counseling, group teaching

SUMMARY:
The investigators will test the hypothesis that a LOW CARB hypocaloric diet will reduce body weight over six months more than a LOW FAT hypocaloric diet. In addition to body weight, the investigators will measure cardiovascular and metabolic variables and will take blood samples in order to determine whether certain metabolites may predict the diet success.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index > 27 kg/m2
* No chronic medication (except oral contraceptives and L-Thyroxine) or possibility to stop medication for study duration
* Able to give written informed consent

Exclusion Criteria:

* Pregnancy and nursing
* Severe cardiovascular, liver, kidney, hepatic or orthopedic disease that need treatment
* Metabolic or endocrine disease that need treatment
* Hypertension blood pressure > 160/95 mmHg or need of > 2 drugs
* Previous stroke or cerebral ischemia
* Significant neurologic or psychiatric disease
* Any kind of eating disorder
* Bariatric surgery in the past
* Drug or alcohol abuse
* Any cancer in the past
* Acute and chronic infections
* Metallic implants (e.g. pace makers) or conditions that do not allow MRI scans
* Body weight > 130 kg

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2007-04; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Body weight reduction | Month 6

SECONDARY OUTCOMES:
Weight maintenance | Month 12 - 36
  follow up assesement after 6 months diet
Reduction of visceral adipose tissue mass | Month 6
Reduction of left ventricular mass | Month 6
Influence on energy expenditure and fat oxidation rates | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Jens Jordan, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Experimental & Clinical Research Center, Berlin, Germany

REFERENCES:
- [Derived] Haufe S, Engeli S, Kaminski J, Witt H, Rein D, Kamlage B, Utz W, Fuhrmann JC, Haas V, Mahler A, Schulz-Menger J, Luft FC, Boschmann M, Jordan J. Branched-chain amino acid catabolism rather than amino acids plasma concentrations is associated with diet-induced changes in insulin resistance in overweight to obese individuals. Nutr Metab Cardiovasc Dis. 2017 Oct;27(10):858-864. doi: 10.1016/j.numecd.2017.07.001. Epub 2017 Jul 11. PMID 28958691
- [Derived] Haufe S, Haas V, Utz W, Birkenfeld AL, Jeran S, Bohnke J, Mahler A, Luft FC, Schulz-Menger J, Boschmann M, Jordan J, Engeli S. Long-lasting improvements in liver fat and metabolism despite body weight regain after dietary weight loss. Diabetes Care. 2013 Nov;36(11):3786-92. doi: 10.2337/dc13-0102. Epub 2013 Aug 20. PMID 23963894
- [Derived] Engeli S, Utz W, Haufe S, Lamounier-Zepter V, Pofahl M, Traber J, Janke J, Luft FC, Boschmann M, Schulz-Menger J, Jordan J. Fatty acid binding protein 4 predicts left ventricular mass and longitudinal function in overweight and obese women. Heart. 2013 Jul;99(13):944-8. doi: 10.1136/heartjnl-2013-303735. Epub 2013 Apr 18. PMID 23598540
- [Derived] Utz W, Engeli S, Haufe S, Kast P, Bohnke J, Haas V, Hermsdorf M, Wiesner S, Pofahl M, Traber J, Luft FC, Boschmann M, Jordan J, Schulz-Menger J. Moderate dietary weight loss reduces myocardial steatosis in obese and overweight women. Int J Cardiol. 2013 Aug 10;167(3):905-9. doi: 10.1016/j.ijcard.2012.03.104. Epub 2012 Apr 10. PMID 22494864
- [Derived] Haufe S, Utz W, Engeli S, Kast P, Bohnke J, Pofahl M, Traber J, Haas V, Hermsdorf M, Mahler A, Busjahn A, Wiesner S, Otto C, Mehling H, Luft FC, Boschmann M, Schulz-Menger J, Jordan J. Left ventricular mass and function with reduced-fat or reduced-carbohydrate hypocaloric diets in overweight and obese subjects. Hypertension. 2012 Jan;59(1):70-5. doi: 10.1161/HYPERTENSIONAHA.111.178616. Epub 2011 Nov 7. PMID 22068866
- [Derived] Utz W, Engeli S, Haufe S, Kast P, Hermsdorf M, Wiesner S, Pofahl M, Traber J, Luft FC, Boschmann M, Schulz-Menger J, Jordan J. Myocardial steatosis, cardiac remodelling and fitness in insulin-sensitive and insulin-resistant obese women. Heart. 2011 Oct;97(19):1585-9. doi: 10.1136/hrt.2011.224451. Epub 2011 Jul 20. PMID 21775510
- [Derived] Haufe S, Engeli S, Kast P, Bohnke J, Utz W, Haas V, Hermsdorf M, Mahler A, Wiesner S, Birkenfeld AL, Sell H, Otto C, Mehling H, Luft FC, Eckel J, Schulz-Menger J, Boschmann M, Jordan J. Randomized comparison of reduced fat and reduced carbohydrate hypocaloric diets on intrahepatic fat in overweight and obese human subjects. Hepatology. 2011 May;53(5):1504-14. doi: 10.1002/hep.24242. Epub 2011 Mar 11. PMID 21400557